CLINICAL TRIAL: NCT02597465
Title: A Randomized, Open-Label, Comparative, Parallel-Group, Multicenter Study of SPARC1507 in Subjects With Cancer
Brief Title: A Randomized, Open-Label, Comparative, Parallel-Group, Multicenter Study of SPARC1507
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided not to initiate the study for alternate commercial strategy
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLR_15_07
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Advanced Biliary Tract Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPARC1507 (Experimental): SPARC1507
  Interventions: Drug: SPARC1507
- Chemotherapy (Experimental): Chemotherapy
  Interventions: Drug: Reference1507

INTERVENTIONS:
Drug: SPARC1507 — The administered dose is calculated based on the BSA calculated for the subject on Day 1 of the Cycle
  Arms: SPARC1507
Drug: Reference1507 — Investigators choice including chemotherapy or supportive therapy
  Arms: Chemotherapy

SUMMARY:
An open label study to determine the efficacy and safety of SPARC1507

DETAILED DESCRIPTION:
Subjects with advanced Biliary tract carcinoma meeting the eligibility criteria will be randomized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of advanced/metastatic biliary tract cancer
* Male or female ≥ 18 years old
* Participants must have measurable disease according to RECIST
* ECOG performance status ≤ 1

Exclusion Criteria:

* Known hypersensitivity to trial treatments, or their excipients
* Prior history of treatment with any taxane therapy
* Cardiovascular disorders as per Investigator's discretion
* The subject has received radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) of subjects treated with SPARC1507 versus IC, per Response Evaluation Criteria in Solid Tumors version 1.1 | 3 years and 6 months

SECONDARY OUTCOMES:
Overall survival in subjects treated with SPARC1507 versus Investigators choice | 3 years and 6 months
Overall response rate in subjects treated with PICN versus Investigators choice | 3 years and 6 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC study site, Aurora, Colorado, United States